CLINICAL TRIAL: NCT00889811
Title: Effect of Lower Limb Remote Preconditioning on Myocardial Injury in Patients Undergoing Off-pump Coronary Artery Bypass Graft Surgery
Brief Title: Effect of Remote Preconditioning in Patients Undergoing Off-pump Coronary Artery Bypass Graft Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Jeon, YunSeok, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: H-0806-060-247
Record Dates: First submitted 2009-04-28; First posted 2009-04-29 (Estimated); Last update posted 2009-10-08 (Estimated); Status verified 2009-10

CONDITIONS: Ischemic Heart Disease
Keywords: OPCAB; RIPC
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: remote ischemic preconditioning — remote ischemic preconditioning (4 x 5 min lower limb ischemia with pneumatic cuff up to 200 mmHg with an intervening 5 min reperfusion; 2 cycles; before and after the coronary anastomosis )
  Other Names: Blood pressure pneumatic cuff

SUMMARY:
In recent several clinical trials, remote preconditioning showed very powerful myocardial protection. However, the myocardial protective effect by remote preconditioning was not evaluated on the patients undergoing off pump coronary artery bypass graft surgery (OPCAB).

The investigators hypothesized that the lower limb remote preconditioning could protect the myocardium during the OPCAB. In this study, the investigators will try to evaluate whether remote preconditioning could induce myocardial protection on the OPCAB patients.

DETAILED DESCRIPTION:
In recent two clinical trials on the patients undergoing cardiac surgery, remote preconditioning showed very powerful myocardial protection by simple and safe procedures such as the brief inflation of pneumatic tourniquet on the upper or lower limb. However, despite these impressive results, the clinical studies are lacking yet. Moreover, two previous studies were done on the cardiac surgery with cardiopulmonary bypass. Considering different mechanism, level of myocardial injury and the increasing popularity of OPCAB, we need the clinical study on remote preconditioning with the OPCAB patients.

In this study, we will conduct randomized controlled clinical trials in which the remote preconditioning was induced by lower limb ischemia with double-blinded technique. Myocardial injury will be assessed by postoperative serum troponin I levels and they will be compared with those of control group.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing elective off pump coronary artery bypass graft surgery

Exclusion Criteria:

* unstable angina
* preoperative use of inotropics or mechanical assist device,
* left ventricular ejection fraction less than 30%,
* major combined operation such as aortic surgery or carotid endarterectomy,
* severe liver, renal and pulmonary disease,
* recent myocardial infarction (within 7 days),
* recent systemic infection or sepsis (within 7 days)
* peripheral vascular disease affecting lower limbs
* amputation of the lower limbs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2009-03; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
postoperative serum troponin I levels | postoperatibe 1, 6, 12, 24, 48, 72 hr

CONTACTS AND LOCATIONS:
Overall Officials: YunSeok Jeon, Professor, Study Director — Department of Anesthesiology and Pain Medicine, SNUH
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Hong DM, Jeon Y, Lee CS, Kim HJ, Lee JM, Bahk JH, Kim KB, Hwang HY. Effects of remote ischemic preconditioning with postconditioning in patients undergoing off-pump coronary artery bypass surgery--randomized controlled trial. Circ J. 2012;76(4):884-90. doi: 10.1253/circj.cj-11-1068. Epub 2012 Feb 3. PMID 22301846